CLINICAL TRIAL: NCT01953432
Title: Pharmacogenetic Trial of Noradrenergic Medication for Treatment of Cocaine Abuse
Brief Title: Pharmacogenetic Trial of Doxazosin for Treatment of Cocaine Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-014-12F; 1IK2CX000946-01 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-10-01 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Cocaine Dependence
Keywords: Cocaine-Related Disorders; Cocaine; Doxazosin; Cardiovascular Agents; Antihypertensive Agents; Adrenergic alpha-1 Receptor Antagonists; Adrenergic alpha-Antagonists; Adrenergic Antagonists; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Therapeutic Uses; Pharmacologic Actions; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Doxazosin; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxazosin (Experimental): Doxazosin is a long-acting and selective alpha 1-NE blocker, which inhibits the binding of norepinephrine to alpha receptors in the autonomic nervous system.
  Interventions: Drug: Doxazosin
- Placebo (Placebo Comparator): Matched placebo daily dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin — Doxazosin is initiated at 2 mg/wk, and titrated up to a maximum of 8 mg/day over approximately 4 weeks. Participants will be maintained on 8mg daily dosing until week 13. The subjects will undergo the discontinuation from the study medication during weeks 14 -15.
  Other Names: Cardura (Doxazosin Mesylate)
  Arms: Doxazosin
Drug: Placebo — Matched placebo daily dosing
  Other Names: Sugar pills (capsule)
  Arms: Placebo

SUMMARY:
Cocaine use disorders affect approximately 1.5 million Americans annually. Currently, there are no US Food and Drug Administration approved medications for treatment of cocaine dependence; however, both animal and human studies suggest that medications affecting the noradrenergic system can reduce cocaine craving and use. The investigators will study the effect of doxazosin, an alpha-1 adrenergic antagonist, in reducing cocaine use and anxiety symptoms among cocaine-dependent individuals. In addition, the investigators will identify genetic subpopulations of participants who preferentially respond to the medication.

DETAILED DESCRIPTION:
The noradrenergic system, especially the alpha 1-adrenergic receptor, may play an important role in cocaine addiction in humans. Doxazosin is a long-acting and selective alpha 1-adrenergic receptor blocker, which inhibits the binding of norepinephrine to alpha receptors in the autonomic nervous system. This study will evaluate the efficacy of doxazosin in reducing cocaine-using behavior in treatment seeking cocaine-dependent individuals, and will guide future pharmacotherapy trials using Doxazosin or related alpha 1 receptor antagonists for treatment of cocaine addiction.

This 12-week double-blind, placebo controlled clinical trial will provide treatment for cocaine-dependent patients and includes a 8-week maintenance medication trial (weeks 3-10). At the end of this period, subjects will have a 2-week study medication taper (weeks 11-12). Qualifying subjects will be randomized to receive Doxazosin up to 8 mg/day or placebo.

At the beginning of week 1, participants will receive Doxazosin, or placebo according to their randomized assignments, and are maintained on these agents through week 12. At the end of the study (weeks 11-12), participants will undergo discontinuation from active/inactive medication over a 2-week period. Subjects who wish to be transferred to an appropriate treatment program or research program will be referred to upon request, during the study weeks 11-12.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and HIPAA authorization form
2. Subject is cooperative, understands the risks and benefits, and is willing and able to adhere to study requirements
3. Any race or ethnic origin
4. Diagnosis of cocaine-dependence according to DSM-IV criteria
5. Between the ages of 18 and 64
6. Must be current users of cocaine with self-reported use of cocaine within the last 90 days, or at least one cocaine-positive urine during screening.
7. Women of childbearing age are eligible to be included in the study if they have a negative pregnancy test at screening, agree to adequate contraception to prevent pregnancy, to have monthly pregnancy tests, and they understand the risk of fetal toxicity due to medication.
8. Must be in good general health as determined by self-report and/or CPRS-based medical history, general clinical examination conducted by a study physician, and lab tests. HIV testing will be recommended but is not required for participation in this study.
9. Motivated to discontinue or reduce cocaine use during the period of the study, as evidenced both by the judgment of the Investigator or designee and by the subject's compliance level with the requirement for attendance at clinic visits, such that weekly urine sample requirements for inclusion criteria are fully met.

Exclusion Criteria:

1. Current diagnosis of other drug dependence, especially alcohol or benzodiazepine dependence, or abuse (other than cocaine, tobacco, or cannabis)
2. Significant medical conditions (e.g., major cardiovascular, renal, endocrine, hepatic disorders) such as abnormal liver function (with laboratory findings of SGOT or SGPT greater than three times normal), hypotension, a current cardiac condition that in the opinion of the investigator would contraindicate Doxasozin treatment, and those having a high risk of cardiovascular disease, seizure disorders, or another significant underlying medical condition which would contraindicate Doxazosin treatment
3. Lifetime schizophrenia, bipolar disorder, or other psychotic disorders (excluding substance-induced psychotic disorders)
4. Actively considering plans of suicidality or homicidality
5. Women planning to become pregnant or breastfeed during the study, refusal to use a reliable form of birth control, or refusal of monthly pregnancy testing
6. Subjects who are prescribed certain anti-hypertension drugs (i.e. doxasozin) will be excluded because these medications may interact with Doxazosin's brain effects in reducing cocaine abuse
7. Subject has participated in another clinical trial or received any other investigational compound within 7 days prior to being randomized into this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl I Shorter, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxazosin: Doxazosin is a long-acting and selective alpha 1-NE blocker, which inhibits the binding of norepinephrine to alpha receptors in the autonomic nervous system.
  Doxazosin (target 8mg/day) Induction - Week 1: 1mg once daily over days 1--3; 2mg once daily over days 4-7; Week 2: 4mg once daily over days 8-10; 8mg once daily over days 11-14; Week 3: 8mg once daily over days 15-end of week 10
  Doxazosin tapered over weeks 11-12 -- Week 11: 4mg on Monday, Tuesday, Wednesday, and Thursday and 1mg for the duration of week 11. During week 12, subjects will receive 1mg on Monday, Tuesday, and Wednesday only. No further medication will be given for the remainder of week 12.
Period: Overall Study
Arm/Group | Doxazosin | Placebo
Started | 22 | 21
Completed | 8 | 6
Not Completed | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxazosin | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 53.4 [26 to 61] | 54.9 [43 to 62] | 54.2 [26 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 17 | 36
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 21 | 43
Lifetime cocaine years [Mean (Full Range); unit: years] | 24.5 [4 to 43] | 24.1 [14 to 38] | 24.3 [4 to 43]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cocaine-positive Urines
Description: Over period of 12 weeks with 43 participants total (Doxazosin group = 22; Placebo group = 21), the overall percentage of cocaine positive urines per treatment group
Time Frame: Up to 12 weeks, or for the duration of the participant's involvement in the study
Population: Study population was comprised of 43 cocaine-dependent individuals who met inclusion criteria for this study.
Measure: Number; unit: percentage of cocaine-positive urines
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 22 | 21
percentage of cocaine-positive urines | 67.6 | 69
Statistical Analysis 1: Comparison: Doxazosin; Test type: Other; Odds Ratio (OR) = 0.75 — Probability of 0.75 that the OR exceeded 1.00 (OR = 1.01, 95% CI = 0.98-1.05)
Statistical Analysis 2: Comparison: Placebo; Test type: Other; Odds Ratio (OR) = 0.96 — Probability of 0.96 that the odds ratio exceeded 1.00 (OR = 1.03, 95% CI = 1.00-1.07)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each visit (Monday, Wednesday, Friday) during the active (medication) portion of the study for each participant (12 weeks).
Arm/Group | Doxazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 8/22 | 5/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxazosin (N=22) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lightheadedness (General disorders) | 1 (1) | 1 (1)
Cold/Viral Illness (Infections and infestations) | 1 (1) | 1 (1)
Stomach Pain/Indigestion (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swelling (Immune system disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergies (Immune system disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Muscle twitching (General disorders) | 0 (0) | 1 (1)
Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Increased Drug Craving (Psychiatric disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a protocol amendment and the primary outcome measure was changed. The planned analysis was revised to a Bayesian approach to ensure more robust analysis of data given smaller sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT01953432/Prot_SAP_000.pdf